CLINICAL TRIAL: NCT01912443
Title: Safety Study of Bevacizumab Plus Chemotherapy To Treat Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Proswell Medical Corporation (Industry)
Responsible Party: Principal Investigator, Ruihua Xu, vice president of SunYat-sen University Cancer Center,head of medical oncology department, Sun Yat-sen University
Other Study IDs: ML28629
Record Dates: First submitted 2013-07-24; First posted 2013-07-31 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bevacizumab Plus Chemotherapy
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — 5 mg/Kg, IV (in the vein) on day 1 and day 14 of each 28 day cycle. Number of Cycles: until progression.
  Other Names: Avastin

SUMMARY:
To assess the safety profile of bevacizumab in combination with chemotherapy for the treatment of metastatic colorectal cancer

DETAILED DESCRIPTION:
This is a multi-centre, observational, non-interventional study. Patients with metastatic colorectal cancer eligible for Bevacizumab in combination with chemotherapy treatment will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* with histologically confirmed metastatic colorectal cancer
* patients with metastatic colorectal cancer who are eligible for Bevacizumab in combination with chemotherapy treatment
* Written informed consent
* Unlimited line of treatment (first-line or second line is not limited)

Exclusion Criteria:

Patients who are not eligible for Bevacizumab treatment according to locally approved Bevacizumab China package insert will be excluded. The following patients are not eligible for Bevacizumab treatment according to local Bevacizumab China package insert:

* Recent history of serious hemorrhage or hemoptysis of ≥1/2 teaspoon of red blood
* Proteinuria at baseline: Patients discovered to have ≥ 2 grams of proteinuria/24 hours *

  * The measurement of 24-hour proteinuria level is recommended for patients with moderate to high proteinuria risk indicated by clinical judgement. The treatment with bevacizumab should be delayed when proteinuria is ≥2g/24 hours.
* Major surgical procedure within 28 days prior to treatment initiation, or not fully healed wounds
* Pregnant or lactating women
* Excluding patients known to be allergic to bevacizumab or any of the excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed metastatic colorectal cancer are eligible
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events of special interest | Four years
  Gastrointestinal perforation, thromboembolic event, wound healing complication, bleeding, hypertension and proteinuria
Incidence, nature and severity of bevacizumab related serious adverse events | Four years
Onset time of adverse event associated with bevacizumab | Four years
Laboratory parameters | Four years
  Complete blood cell count, electrolytes, hepatic and renal function, coagulation parameters, urinalysis or urine protein

SECONDARY OUTCOMES:
Overall survival (OS) | Four years
  Time from the diagnosis of colorectal cancer to death due to various causes. Patients who do not die at the end of study will be truncated when they do not die at the last collection.
Overall response rate (ORR) of treatment line | Four years
  The best overall response status determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria is defined as the best response status recorded from the enrollment to disease progression (the minimal measurement from baseline assessment is used as the reference for progression). ORR includes complete response (CR) and partial response (PR). The value of change will be summarized according to different treatment lines.
Progression-free survival (PFS) of treatment line: | Four years
  Time from the enrollment to disease progression or death due to various causes, whichever is earlier (Disease progression is according to RECIST 1.1 criteria for tumor assessment). Patients who do not have disease progression or death at the end of study will be truncated at the last tumor assessment. The value of change will be summarized according to different treatment lines.
One-year disease-free progression rate of treatment line | One year
  The proportion of patients without disease progression within one year since enrollment or with death for other reasons based on analytical population. The value of change will be summarized according to different treatment lines.
One-year survival rate of treatment line | One year
  The proportion of patients without death within one year since enrollment based on analytical population. The value of change will be summarized according to different treatment lines.
Overall survival (OS) of treatment line | Four years
  Time from the enrollment to death due to various causes. Patients who do not die at the end of study will be truncated when they do not die at the last collection.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Liaoning Cancer Hosptial & Institute, Shenyang, Liaoning
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan
  - First Affiliated Hospital of PLA General Hospital, Beijing
  - Chinese PLA General Hospital, Beijing